CLINICAL TRIAL: NCT06676826
Title: Treatment of Periodontal Intra-bony Defects With a Volume Stable Collagen Matrix or Deproteinized Bovine Bone Mineral With 10% Collagen. A 12-month Multi-center Randomized Controlled Trial
Brief Title: Treatment of Periodontal Intra-bony Defects With a Volume Stable Collagen Matrix or Deproteinized Bovine Bone Mineral With 10% Collagen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-D0026
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (VCMX) (Experimental): The periodontal infrabony defect will be opened by a papilla preservation flap, the root surface will be thoroughly cleaned with hand instruments and ultrasonic scalers, then the bony defect will be filled with a volume-stable collagen matrix (VCMX) only.
  Interventions: Device: Infrabony defects will be filled with a volume-stable collagen matrix (VCMX)
- Control Group (Deproteinized bovine bone mineral) (Active Comparator): The periodontal infrabony defect will be opened by a flap, the root surface will be thoroughly cleaned with hand instruments and ultrasonic scalers, then the bony defect will be filled with deproteinized bovine bone mineral with 10% collagen.
  Interventions: Device: Infrabony defects will be filled treated with a deproteinized bovine bone mineral with 10% collagen

INTERVENTIONS:
Device: Infrabony defects will be filled with a volume-stable collagen matrix (VCMX) — Infrabony defects will be filled with a volume-stable collagen matrix
  Other Names: VCMX
  Arms: Test Group (VCMX)
Device: Infrabony defects will be filled treated with a deproteinized bovine bone mineral with 10% collagen — Infrabony defects will be filled with with a deproteinized bovine bone mineral with 10% collagen
  Other Names: DBBM
  Arms: Control Group (Deproteinized bovine bone mineral)

SUMMARY:
To compare the healing of intrabony periodontal defects treated with either open flap debridement and a volume-stable collagen matrix (VCMX) or a deproteinized bovine bone mineral with 10% collagen. The results will shed light on the clinical potential of VCMX in regenerative periodontal surgery and help to develop new treatment strategies.

ELIGIBILITY:
Inclusion Criteria

* Patients with localized or generalized periodontitis Stage III and Stage IV, Grade A-B-C
* Males and females
* Age at least 18 years and older
* Presence of interdental intra-bony defects (I, II and III walls) in either the maxilla or the mandible with a PD ≥ 6 mm
* Defects with an intra-bony component > 3 mm for both groups
* Intra-bony defect located only at one aspect (mesial or distal)
* Presence of at least 2 mm of keratinized soft tissue. Exclusion Criteria
* Patients with systemic disease that could interfere with periodontal wound healing
* Prolonged antibiotic treatment or anti-inflammatory treatment within 4 weeks prior to surgery
* Pregnant or lactating
* Smokers with > 10 cig./day
* Patients with FMPS and FMBS > 25 % after completion of non-surgical periodontal therapy
* Multi-rooted teeth with furcation involvement
* Third molars
* Teeth with circumferential defects
* Interdental craters
* Written Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) change | 12 months
  Clinical attachment level (CAL) change in mm: the distance from the cemento-enamel junction to the bottom of the clinical periodontal pocket is being measured

SECONDARY OUTCOMES:
Microbiological analysis | 1, 3, 12 weeks
  Quantification of the concentration of host-derived biomarkers (interleukin-1beta (IL-1b), IL-10, matrix-metalloproteinase- 8(MMP-8)) and periodontal bacterial species by means of gingival crevicular fluid and the biofilm sampling
Bleeding on probing (BoP) | Baseline, 12 months
  Assessment of number of bleeding spots (percentage 0-100%) upon gentle probing of PPD at each test and control tooth site
Pocket probing depth (PPD) | Baseline, 12 months
  With a periodontal probe with mm markings, the distance between the gingival margin and the bottom of the pocket will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Stähli, MD, Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No